CLINICAL TRIAL: NCT04775407
Title: COVID-19 Serological Testing of Patients With a Diagnosis of Schizophrenia, Schizoaffective Disorder or Bipolar Affective Disorder From the Catchment Area of the Capital Region of Denmark
Brief Title: COVID-19 Serological Testing of Patients With a Mental Disorder From the Catchment Area of the Capital Region of Denmark
Status: Terminated | Type: Observational
Why Stopped: Due to the development of the pandemic
Sponsor: Anders Fink-Jensen, MD, DMSci (Other)
Responsible Party: Sponsor-Investigator, Anders Fink-Jensen, MD, DMSci, MD Proffessor, Psychiatric Centre Rigshospitalet
Organization: Psychiatric Centre Rigshospitalet (Other)
Other Study IDs: COVID-19 RHP
Record Dates: First submitted 2021-02-22; First posted 2021-03-01 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Covid19; Severe Mental Disorder
MeSH Terms: conditions — COVID-19; Mental Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sampling for SARS-CoV-2 antibodies analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screening: Serological SARS-CoV-2 test
  Interventions: Procedure: blood sampling

INTERVENTIONS:
Procedure: blood sampling — IgM og IgG analysis

SUMMARY:
The pandemic of coronavirus disease 2019 (COVID-19) caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has lately caused worldwide health problems. Patients suffering from a severe mental disorder are at increased risk for infectious diseases. The primary aim of the present surveillance study is to perform COVID-19 serological testing on patients with a diagnosis of schizophrenia, schizoaffective disorder or a bipolar affective disorder. Patients from the catchment area of the Capital Region of Denmark will be COVID-19 tested at baseline (0 months) and again at 6 and 12 months, in order to follow the spread of COVID-19 among this vulnerable patient population.

DETAILED DESCRIPTION:
Patients suffering from severe mental illness could be in increased risk for a severe outcome if infected with COVID-19. Also, there are reports on fewer treatment activities among psychiatric patients (e.g. higher heart disease mortality), lower hospitalization rate and fewer invasive cardiac procedures among persons with schizophrenia than among the general population. This conveys a risk not only for the patient but for the spread of COVID-19 in the community. At present, we expect the outcome of a COVID-19 infection to be worse among the mentioned psychiatric patient population, but whether the spread of COVID-19 differs from the pattern observed in the general population is unknown. This information is of pivotal interest to come up with sufficient treatment strategies - especially when facing a possible second surge in the COVID-19 spread. Moreover, it is to the best of our knowledge unknown whether a possible CNS COVID-19 infection will worsen existing psychopathology among patients with severe schizophrenia, schizoaffective- or bipolar affective disorder. The study is exploratory in nature including as many patients as possible for testing. The target population is patients diagnosed with schizophrenia, schizoaffective disorder or a bipolar affective disorder receiving in-patient or out-patient care via one of the psychiatric centres in The Mental Health Services in the Capital Region of Denmark. Each patient will attend 3 study visits during a period of 12 months. A blood sample for IgG and IgM analysis for will be drawn at every visit.

ELIGIBILITY:
Inclusion Criteria:

1. Informed oral and written consent
2. Age ≥ 18 years
3. Patients with a diagnosis of schizophrenia, schizoaffective disorder or a bipolar affective disorder, according to the criteria of ICD10 (International Classification of Diseases, World Health Organization (WHO))
4. Receiving psychiatric treatment from a hospital in- or outpatient-clinic in the catchment area of the Capital Region of Denmark

Exclusion Criteria:

1. Patient with signs of infection should initially be transferred to the national test centres antigen-PCR testing. These patients will be offered to participate in next blood sampling interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is patients diagnosed with schizophrenia, schizoaffective disorder or a bipolar affective disorder receiving in-patient or out-patient care via one of the psychiatric centres in The Mental Health Services in the Capital Region of Denmark
Sampling Method: Non-Probability Sample
Enrollment: 1355 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
The incidence of positive serological COVID-19 test result | 18 month
  A blood sample from each patient is analyzed for COVID-19 antibodies

SECONDARY OUTCOMES:
Registered death (number), hospital admissions (number), changes in out-patients clinic contacts (number), changes in suicidal behavior (score on medical scale) and changes in psychopharmacological treatment (registered changed in medial journal). | 18 month
  Data from Danish registers and from patient medical records are correlated with the possible presence of COVID-19 antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric Centre Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sass MR, Juul TS, Skov R, Iversen K, Harritshoj LH, Sorensen E, Ostrowski SR, Andersen O, Ekstrom CT, Ullum H, Nielsen J, Hageman I, Fink-Jensen A. SARS-CoV-2 seroprevalence among patients with severe mental illness: A cross-sectional study. PLoS One. 2022 Mar 1;17(3):e0264325. doi: 10.1371/journal.pone.0264325. eCollection 2022. PMID 35231037